CLINICAL TRIAL: NCT02937961
Title: Early Versus Late Sustained Low Efficiency Dialysis in Critically Ill Cirrhotics With Septic Shock and Acute Kidney Injury -A Pilot Randomized Controlled Trial
Brief Title: Early Versus Late Sustained Low Efficiency Dialysis in Critically Ill Cirrhotics With Septic Shock and Acute Kidney Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Septic Shock-001
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-01

CONDITIONS: Cirrhotics With Septic Shock and Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early SLED (Experimental)
  Interventions: Biological: Early SLED
- Late SLED (Active Comparator)
  Interventions: Biological: Late SLED

INTERVENTIONS:
Biological: Early SLED — withing 6 to 12 hours
  Arms: Early SLED
Biological: Late SLED — when absolute indications will meet
  Arms: Late SLED

SUMMARY:
Consecutive patients with cirrhosis and septic shock with AKI who give written informed consent will be included in this prospective trial. At baseline NT-Pro BNP, urine N-GAL will be done for all patients. A baseline serum blood sample (10 ml) and urine sample will be stored. Septic shock will be defined by the presence of two or more diagnostic criteria for the systemic inflammatory response syndrome, proven or suspected infection with hypotension non-responsive to adequate fluid resuscitation assessed by no evidence of stroke volume variation on flow track and need of a vasopressor to achieve a target mean arterial pressure (MAP) of ≥ 65 mm Hg. A record of CVP, IVC diameter and B-lines on ultrasound lung would also be done. Patients with age less than 18 years, severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD) pregnancy, chronic kidney disease on hemodialysis, patients already meeting emergency criteria for immediate hemodialysis at the time of randomization as specified in the late group, patients transferred from other hospitals who have already been on hemodialysis before their arrival in the intensive care unit, extremely moribund patients with an expected life expectancy of less than 24 hours, failure to give informed consent from family members.

ELIGIBILITY:
Inclusion Criteria:

- Patients with Cirrhosis with septic shock associated AKI (Acute Kidney Injury) stage 3 AKIN/KDIGO stage 2.

Exclusion Criteria:

* Patients with age less than 18 years
* Severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, Coronary Obstructive Pulmonary Disease)
* Pregnancy
* Chronic kidney disease on hemodialysis
* Patients with Hepatorenal Syndrome, post renal obstructive AKI, AKI due to suspected based on history,urinalysis and past clinical records-glomerulonephritis, interstitial nephritis or vasculitis
* Patients already meeting emergency criteria for immediate hemodialysis at the time of randomization as specified in the late group (serum potassium>6 meq/lt, metabolic acidosis ph<7.12, acute pulmonary edema, severe volume overload with hypoxemia non-responsive to diuretic treatment)
* Patients transferred from other hospitals who have already been on hemodialysis before their arrival in the intensive care unit
* Extremely moribund patients with an expected life expectancy of less than 24 hours
* Failure to give informed consent from family members.
* Hemodynamic instability requiring very high dose of vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival in both groups | 28 days

SECONDARY OUTCOMES:
Incidence of intradialytic hypotension in both groups | 48 hours
Hemodynamic stability in both groups | 48 hours
Dialysis efficiency as measured by Urea Reduction ratio in both groups | 2 days
Achievement of target ultrafiltration goals in both groups | 48 hours
Recovery in renal functions in both groups | 14 days
  Recovery is defined as an increase in urine output to more than 400 ml/day
Duration of Intensive Care Unit stay in both groups | 28 days
Duration of mechanical ventilation in both groups | 28 days
Improvement in Sequential Organ Failure Assessment ( by 2 points) scores in both groups | 28 days
Improvement in SOFA, Model for End stage Liver Disease ( by 2 points) scores | 28 days
Improvement in Acute Physiology and Chronic Health Evaluation ( by 2 points) scores | 28 days
Improvement in lactic acidosis and lactate clearance at 6 initiation of dialysis in both groups | 6 hours
Improvement in lactic acidosis and lactate clearance at 24 hours after initiation of dialysis in both groups | 12 hours
Improvement in lactic acidosis and lactate clearance at 24 hours after initiation of dialysis in both groups | 24 hours
Death related with renal failure in both groups | 7 day
Mortality due to renal failure related in both groups. | 7 day

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maiwall R, Pasupuleti SSR, Agarwal P, Thomas S, Tevethia HV, Mathur RP, Sarin SK. Early Versus Late Dialysis in Cirrhosis Patients and Septic Shock (ELDICS Study): A Randomized Controlled Trial (NCT02937961). JGH Open. 2025 Sep 24;9(9):e70216. doi: 10.1002/jgh3.70216. eCollection 2025 Sep. PMID 41020192
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787